CLINICAL TRIAL: NCT00828399
Title: Efficacy of Glutamine in the Prevention of Acute Radiation Enteritis Among Patients Treated With Radiation of Abdomen and Pelvis.
Brief Title: Prevention of Acute Radiation Enteritis With Glutamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Castilla-León Health Service (Other)
Responsible Party: MD Alfonso Vidal Casariego, Complejo Asistencial de Leóm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 001-2008-BecaSacyl
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2009-01

CONDITIONS: Acute Radiation Enteritis
Keywords: Radiotherapy; Diarrhoea; Glutamine; Oxydative stress; Calprotectin; Citrulline
MeSH Terms: conditions — Diarrhea | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Experimental)
  Interventions: Dietary Supplement: Glutamine
- Whole protein (Placebo Comparator)
  Interventions: Dietary Supplement: Whole protein

INTERVENTIONS:
Dietary Supplement: Glutamine — Oral glutamine 30g/day
  Arms: Glutamine
Dietary Supplement: Whole protein — Oral whole protein 30 g/day
  Arms: Whole protein

SUMMARY:
Ionizing radiation has cytotoxic effects, and is commonly used as treatment for neoplasm. A common adverse effect of radiation is acute diarrhoea. Glutamine is an aminoacid with antioxidant effects that can protect tissues of damage dued to radiation. The investigators designed a randomized, double-blind trial phase III to study if glutamine prevents acute radiation enteritis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yr
* Gynaecological,prostatic, rectal or other abdominal cancer
* Radiotherapy with/without chemotherapy

Exclusion Criteria:

* life expectancy < 1 yr
* Age < 18 yr
* gut diseases: inflammatory bowel disease,sprue, irritable bowel disease...
* moderate to severe chronic renal failure
* hepatic cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with acute radiation enteritis | 2 months
  RTOG criteria

SECONDARY OUTCOMES:
Reduction in inflammatory markers and oxydative stress | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Vidal Casariego, MD, Principal Investigator — Sección de Endocrinología y Nutrición. Complejo Asistencial de León
Locations (1):
- Complejo Asistencial de León., León, Leon, Spain

REFERENCES:
- [Result] Kozelsky TF, Meyers GE, Sloan JA, Shanahan TG, Dick SJ, Moore RL, Engeler GP, Frank AR, McKone TK, Urias RE, Pilepich MV, Novotny PJ, Martenson JA; North Central Cancer Treatment Group. Phase III double-blind study of glutamine versus placebo for the prevention of acute diarrhea in patients receiving pelvic radiation therapy. J Clin Oncol. 2003 May 1;21(9):1669-74. doi: 10.1200/JCO.2003.05.060. PMID 12721240
- [Result] Giris M, Erbil Y, Oztezcan S, Olgac V, Barbaros U, Deveci U, Kirgiz B, Uysal M, Toker GA. The effect of heme oxygenase-1 induction by glutamine on radiation-induced intestinal damage: the effect of heme oxygenase-1 on radiation enteritis. Am J Surg. 2006 Apr;191(4):503-9. doi: 10.1016/j.amjsurg.2005.11.004. PMID 16531144
- [Result] Ersin S, Tuncyurek P, Esassolak M, Alkanat M, Buke C, Yilmaz M, Telefoncu A, Kose T. The prophylactic and therapeutic effects of glutamine- and arginine-enriched diets on radiation-induced enteritis in rats. J Surg Res. 2000 Apr;89(2):121-5. doi: 10.1006/jsre.1999.5808. PMID 10729239
- [Result] de Urbina JJ, Jorquera F, Culebras JM, Villares C, Gonzalez-Gallego J, Tunon MJ. Effects of parenteral nutrition supplemented with alanyl-glutamine on nutrition status in rats. JPEN J Parenter Enteral Nutr. 2005 Jul-Aug;29(4):262-5. doi: 10.1177/0148607105029004262. PMID 15961682